CLINICAL TRIAL: NCT07122843
Title: Real Time Guided Meditations for Pain in Virtual Reality Study
Brief Title: VR AI Meditation for Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Almario (Other)
Responsible Party: Sponsor-Investigator, Christopher Almario, Associate Professor of Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004263
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Pain and Anxiety
Keywords: Virtual Reality; Meditation; Guided Meditation
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- VR Guided Meditation (Experimental): Patients will wear a VR headset for approximately 15 minutes. The headset fully covers the eyes, immersing users in a calming, 3D virtual environment. Once the headset is on, patients will engage in a guided meditation experience, set in a nature-themed scene of their choice; options include a lake, beach, mountains, desert, forest, space, and more. An AI-powered guide will lead the meditation, offering real-time, personalized support based on the patient's age and the pain-related information provided during the hospital intake process. The AI is designed to promote relaxation by helping patients focus, breathe deeply, and feel more at ease. The intervention will be standardized for all participants, with each receiving the same duration of exposure in the VR headset and access to an identical selection of nature scenes. The patients will fill our pre and post intervention pain and anxiety surveys. The pre and post surveys will take between 5-10 minutes each to complete.
  Interventions: Device: VR Guided Meditation

INTERVENTIONS:
Device: VR Guided Meditation — Patients will wear a VR headset for approximately 15 minutes. The headset fully covers the eyes, immersing users in a calming, 3D virtual environment. Once the headset is on, patients will engage in a guided meditation experience, set in a nature-themed scene of their choice; options include a lake, beach, mountains, desert, forest, space, and more. An AI-powered guide will lead the meditation, offering real-time, personalized support based on the patient's age and the pain-related information provided during the hospital intake process. The AI is designed to promote relaxation by helping patients focus, breathe deeply, and feel more at ease. The intervention will be standardized for all participants, with each receiving the same duration of exposure in the VR headset and access to an identical selection of nature scenes. The patients will fill our pre and post intervention pain and anxiety surveys. The pre and post surveys will take between 5-10 minutes each to complete.

SUMMARY:
This study aims to assess changes in pain and anxiety as reported by the Pain Numeric Rating Scale (PNRS) and the State-Trait Anxiety Inventory 6 (STAI-6), pre and post a guided meditation in Virtual reality. Objectives of the study are also to determine the feasibility, and patient acceptance of utilizing a LLM-generated guided meditation in VR. Our goal is to learn about any limitations of our approach and provide a pathway for future improvements in creating a VR AI therapist that is optimally aligned with the needs of users.

DETAILED DESCRIPTION:
38 individuals who are admitted to CSMC, who have completed Inpatient Pain Service Center intake form, and who have a baseline pain score of 4 on the PNRS or greater to experience VR guided meditation will be invited to join the study. Patients must have a minimum baseline pain score of 4 or higher on the PNRS to be eligible for evaluation in this study because if a patient begins with no or minimal pain, there is no opportunity for the VR meditation program to produce a measurable reduction in pain levels. Patients will wear a VR headset for approximately 15 minutes. The headset fully covers the eyes, immersing users in a calming, 3D virtual environment. Once the headset is on, patients will engage in a guided meditation experience, set in a nature-themed scene of their choice; options include a lake, beach, mountains, desert, forest, space, and more. An AI-powered guide will lead the meditation, offering real-time, personalized support based on the patient's age and the pain-related information provided during the hospital intake process. The AI is designed to promote relaxation by helping patients focus, breathe deeply, and feel more at ease. The intervention will be standardized for all participants, with each receiving the same duration of exposure in the VR headset and access to an identical selection of nature scenes. Participants will complete pre-intervention pain and anxiety surveys which will take 5-10 minutes followed by a 15-minute experience in VR and we will end with a post-intervention pain (PNRS) and anxiety (STAI-6) surveys (5-10 minutes). The total session will range from 25-35 minutes in length. The study is also determine the feasibility, and patient acceptance of utilizing a LLM-generated guided meditation in VR. The goal is to learn about any limitations of our approach and provide a pathway for future improvements in creating a VR AI therapist that is optimally aligned with the needs of users.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Individuals who are admitted to CSMC and who have completed the Inpatient Pain Service Center intake form.
* Participants must speak one of the program's supported languages (currently English and Spanish)
* Minimum pain score of 4 out 10 on baseline pain survey

Exclusion Criteria:

* Unwilling and/or unable to participate
* Does not understand English or Spanish
* Self-reported history of severe motion sickness
* The presence of a facial/head deformity that will prohibit the wearing of a VR HMD
* Those that require corrective lenses -2.5 or stronger that cannot be corrected with contact lenses
* Legally deaf
* Having had a seizure in the past year
* Unable to understand the instructions or to consent to participation in the study
* Those who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Pain Numeric Rating Scale Pre and Post VR Guided Meditation | Pre VR Use (Baseline) and Post VR Use (after a 15 minutes experience in VR)
  To evaluate impact to pain levels after VR guided meditation (1 time). We will use a validated pain survey and look at Pain Numeric Rating Scale (pre compared to post-VR).

SECONDARY OUTCOMES:
STAI-6 Scores Pre and Post VR Guided Meditation | Pre VR use (Baseline) and Post VR use (after 15-minute experience in VR)
  To evaluate anxiety scores pre and post VR guided meditation on the STAI-6.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher V Almario, MD, MSHPM, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States